CLINICAL TRIAL: NCT00896077
Title: A Safety, Tolerability and Bioavailability Study of Lisofylline After Continuous Subcutaneous (12 mg/kg) and Intravenous (12 mg/kg) Administration in Healthy Subjects and in Subjects With Type 1 Diabetes Mellitus
Brief Title: Subcutaneous Administration of Lisofylline to Healthy Normal Subjects and Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DiaKine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DT-002
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Healthy; Type 1 Diabetes
Keywords: healthy subjects
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — lisofylline

ARMS (2):
- Subcutaneous (Active Comparator): Subcutaneous administration of LSF
  Interventions: Drug: Lisofylline
- IV (Active Comparator): IV administration arm
  Interventions: Drug: Lisofylline

INTERVENTIONS:
Drug: Lisofylline — Lisofylline via i.v. administration vs Lisofylline vs s.c. administration

SUMMARY:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease. Autoimmune diseases happen when the immune system does not identify part of the body as belonging to it. The immune system then destroys that part as if it were an unknown tissue in the body. In T1DM, the body kills the cells in the pancreas that produce insulin. Insulin is the hormone that "unlocks" the cells of the body. It allows glucose to enter and fuel them. Special cells in the body called islets make the insulin. Since glucose cannot enter the cells, it builds up in the blood. The body's cells literally starve to death. Children are at risk of developing T1DM and the risk is much higher than other severe, chronic childhood diseases. The only treatments are a careful diet, planned physical activity, and testing blood sugar levels several times a day. The patient must also inject insulin each day or use an insulin pump. There is no cure for T1DM. Insulin injections are considered life support, because going without insulin for just a few days causes the blood to have too much acid in it and that can lead to death. On the other hand, taking too much insulin makes blood sugar levels go too low, and if untreated, can lead to death as well.

DiaKine is developing Lisofylline to treat the failed immune system. This is what caused T1DM in the first place and it does not go away. The purpose of this study is to see how safe the study drug is. The study is also going to compare the levels of study drug in the blood and to measure the effect of the study drug on other substances in the blood that are linked to type 1 diabetes. These levels will be measured after the study drug is given as an injection under the skin and an injection into the vein. To date, Lisofylline has been tested when given as an injection in the vein.

The investigators hypothesize that Lisofylline will be safe when given as an injection under the skin and in the vein and that levels of study drug will be very similar when given as an injection under the skin and in the vein.

The investigators also hypothesize that Lisofylline will have a positive effect on the substances in the blood that are linked to type 1 diabetes.

DETAILED DESCRIPTION:
Compound: Lisofylline

Protocol Number and Title: DT-002: A Safety, Tolerability and Bioavailability Study of Lisofylline After Continuous Subcutaneous (12 mg/kg) and Intravenous (12 mg/kg) Administration in Healthy Subjects and in Subjects With Type 1 Diabetes Mellitus

Clinical Trial Phase: Phase 1 / Phase 2A

Study Objectives: The primary objective of this study is to assess safety and tolerability of Lisofylline (LSF) in healthy adult subjects and in adult subjects with type 1 diabetes mellitus (DM) following a single dose of LSF 12 mg/kg administered as a continuous subcutaneous (s.c.) infusion over 24 hours, versus a single dose of LSF 12 mg/kg administered as a continuous intravenous (i.v.) infusion over 24 hours.

The secondary objectives of this study are (1) to determine the bioavailability of a single dose of LSF 12 mg/kg administered as a continuous s.c. infusion over 24 hours compared to that of a single dose of LSF 12 mg/kg administered as a continuous i.v. infusion over 24 hours; and (2) an exploratory evaluation of the early efficacy of LSF based upon evaluation of pharmacodynamic (PD) data.

Principal Investigator and Study Site:

Benno G. Roesch, MD Advanced Biomedical Research, Inc. Clinical Research Center 241 Main Street Hackensack, New Jersey 07601 USA

Number of Subjects and Subject Population:

Up to 8 male or female subjects (up to 4 healthy adult male or female subjects and up to 4 male or female subjects with type 1 DM) will be enrolled as two separate cohorts into the study to ensure a total of at least 6 evaluable subjects.

Healthy male or female subjects between 18-45 years of age, inclusive, and male or female subjects, 18-45 years of age, inclusive, with a clinical diagnosis of type 1 DM for a minimum of 2 years, requiring treatment with insulin, and no other clinically significant exclusionary disease or conditions, are eligible to participate in the study.

Study Design: This is an open-label, single-dose, randomized, two-period, two-treatment, crossover study in healthy subjects and in subjects with type 1 DM.

Eligible subjects will be admitted to the Clinic the evening prior to dosing (Day -1, Day 6) during each treatment period, receive their assigned dose of study drug on Day 1 and Day 7, and will remain confined to the Clinic until approximately 48 h following the start of study drug administration (Day 3, Day 9). A washout period of three days will separate the two treatment periods. All subjects will receive a single dose of LSF 12 mg/kg administered via continuous i.v. infusion over a 24-hour period during one treatment period and a single dose of LSF 12 mg/kg administered via continuous s.c. infusion over a 24-hour period during the alternate treatment period.

Healthy subjects and subjects with type 1 DM will comprise two separate cohorts. All subjects will be assigned a treatment sequence according to a randomization schedule that will balance sequence assignments within the two cohorts.

Study Duration: The overall duration of the study for each subject is approximately 30 days. This includes a 21-day screening period, two active treatment periods of three days each separated by a 3-day washout period.

Study Drug: The drug product, LSF for injection, will be supplied by the Sponsor or designee as a 120 mg/mL sterile solution (600 mg LSF/5 mL) in USP type 1 molded clear glass vials. Each subject will receive a single dose of LSF 12 mg/kg as a continuous s.c. infusion over 24 hours during one period, and a single dose of LSF 12 mg/kg as a continuous i.v. infusion over 24 hours during the alternate period in a randomized fashion.

Treatment Groups: There will be two treatment groups: LSF 12 mg/kg as a continuous s.c. infusion over 24 hours and LSF 12 mg/kg as a continuous i.v. infusion over 24 hours.

Study Procedures: After providing written informed consent, subjects will undergo a complete medical history, medication history, physical examination, vital signs evaluation, resting 12 lead electrocardiogram (ECG), clinical laboratory tests [chemistry, hematology, urinalysis, HIV, Hepatitis B & C diagnostic profile and urine drug, alcohol and pregnancy (females only) screen,] within 21 days prior to receiving the first dose of study drug.

On Days 1 and 7, eligible subjects will receive a single dose of LSF 12 mg/kg administered via continuous i.v. infusion over a 24-hour period during one treatment period and a single dose of LSF 12 mg/kg administered via continuous s.c. infusion over a 24-hour period during the alternate treatment period.

Seated blood pressure and pulse rate will be measured on Days 1-3 and 7-9 within 15 min prior to the start of infusion and 1, 4, 12, 24, 36 and 48 h following the start of infusion. A resting 12-lead ECG will be performed on Days 1-2 and Days 7-8 at 1, 8 and 24 h following the start of infusion, and prior to discharge from the Clinic on Day 9. An abbreviated physical examination will be performed on Day 3, prior to discharge from the Clinic and a complete physical examination will be performed on Day 9, prior to discharge from the study. Adverse events (AEs) will be monitored by nursing and medical observations and spontaneous reporting throughout the study. In addition, skin irritation assessments will be performed on Days 1-2 and Days 7-8 within 15 min prior to the start of infusion and 2, 4, 8, 12 and 24 h following the start of infusion.

Blood will be collected for determination of plasma LSF concentration on Days 1-2 and Days 7-8 within 0.5 h prior to the start of infusion (time 0) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18 and 24 h following the start of infusion. On Day 2 and Day 8, blood samples will be collected 5, 10, 15 and 30 min and 1, 2, 3, 4, 6, 8, 10, 12 and 16 h following completion of the 24-h infusion period.

Blood will be collected for evaluation of cytokine, chemokine, insulin and free fatty acid (FFA) serum levels, and for evaluation of STAT4 phosphorylation status of monocytes, on Days 1-2 and Days 7-8 within 0.5 h prior to the start of infusion (time 0) and 24 h following the start of infusion.

Study Endpoints Plasma LSF concentrations and PK assessments: Blood will be collected for determination of plasma LSF concentration at time points noted previously. PK parameters will include AUC0-t, AUC0-inf, Cmax, Tmax, t1/2, kel, CL, Vdss and F.

PD assessments: Blood will be collected for determination of serum cytokine, chemokine, insulin and FFA levels at time points noted previously.

Safety outcome measures: Safety will be based on AEs, vital signs assessments, resting 12-lead ECG evaluations, physical examination findings and clinical laboratory test results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are eligible for participation in the healthy subject cohort of the study:

  1. Ability to understand and provide written informed consent;
  2. Ability to complete the study in compliance with the protocol;
  3. Healthy male or female between 18 and 45 years of age, inclusive;
  4. Female subjects must be non-pregnant and non-lactating and must be surgically sterile, postmenopausal, or willing to use adequate contraception, including but not limited to hormonal contraceptive, diaphragm, condom or intrauterine device, during the course of the study. Female subjects must agree not to attempt to become pregnant during the study;
  5. Male subjects must be willing to use effective birth control if their female partners are of child-bearing potential starting the day prior to the first dose of study drug until the end of the study;
  6. Weigh at least 50 kg (110 lbs);
  7. Body mass Index (BMI) between 19 and 34.5 kg/m2, inclusive;
  8. No clinically significant abnormal findings on the physical examination, medical history, vital signs assessment, resting 12-lead ECG evaluation or clinical laboratory test results during screening;
  9. A negative hepatitis B surface antigen, hepatitis C antibody or HIV antibody test result at screening or within the previous 3 months.
* Subjects who meet all of the following criteria are eligible for participation in the type 1 DM cohort of the study:

  1. Ability to understand and provide written informed consent;
  2. Ability to complete the study in compliance with the protocol;
  3. Male or female between 18 and 45 years of age, inclusive;
  4. If the subject is female, she must be non-pregnant and non-lactating and must be surgically sterile, postmenopausal, or willing to use adequate contraception, including but not limited to hormonal contraceptive, diaphragm, condom or intrauterine device, during the course of the study. Female subjects must agree not to attempt to become pregnant during the study;
  5. Male subjects must be willing to use effective birth control if their female partners are of child-bearing potential starting the day prior to administration of the first dose of study drug until the end of the study;
  6. Weigh at least 50 kg (110 lbs);
  7. Body Mass Index (BMI) between 19 and 34.5 kg/m2, inclusive;
  8. Clinical diagnosis of type 1 DM at least 2 years prior to screening;
  9. Treatment with insulin for at least 1 year and on a stable dose for at least 3 months prior to screening. Dose must be ≤ 0.8 units/kg/day;
  10. Currently self-monitoring blood glucose levels at least daily;
  11. HbA1c level 6-10%, inclusive;
  12. Serum C-peptide level ≤ 0.6 ng/mL;
  13. Serum creatinine < 1.5 mg/dL for males, and <1.4 mg/dL for females;

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from participation in the healthy subject cohort of the study:

  1. A clinically significant laboratory abnormality or other clinical findings indicative of a clinically significant exclusionary disease (including but not limited to renal, hepatic, gastrointestinal, cardiovascular, neurological disease);
  2. History of any significant drug allergy;
  3. History of difficulty with phlebotomy;
  4. Use of any recreational drugs within the past year or a previous history of drug or alcohol abuse;
  5. Positive results from a urine screen for alcohol or substances of abuse at screening or upon admission to the Clinic;
  6. Current smoker or user of any tobacco products;
  7. Use of any prescription drug therapy within 14 days prior to receiving study drug;
  8. Use of any over-the-counter (OTC) drugs or herbal preparations within 72 hours prior to receiving study drug;
  9. Consumption of any caffeine-containing foods or beverages within 24 hours prior to receiving study drug;
  10. Consumption of alcohol within 24 hours prior to admission to the Clinic;
  11. Consumption of any grapefruit or grapefruit-containing juices within 72 hours prior to receiving study drug;
  12. Use of an investigational drug or product, or participation in a drug research study within 30 days prior to receiving drug;
  13. Prior exposure to lisofylline;
  14. The donation of blood (1 pint or more) within 30 days or plasma within 7 days of receiving study drug;
  15. Any condition which in the opinion of Investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he or she took part in the trial
* Subjects meeting any of the following criteria will be excluded from participation in the type 1 DM cohort of the study:

  1. Known or suspected history of significant gastrointestinal, liver or cardiac disease, including stroke, peripheral vascular disease or any related symptom
  2. History of peptic ulcer disease and or gastrointestinal bleeding/perforation;
  3. History or presence of proliferative retinopathy, severe non-proliferative retinopathy, macular edema or presence of untreated diabetic eye disease;
  4. History of treated peripheral or autonomic neuropathy;
  5. History of hypoglycemia unawareness, and/or episodes of severe hypoglycemia within 60 days prior to screening;
  6. Non-healed diabetic ulcer;
  7. Diagnosis of type 2 DM, based upon subject report;
  8. Use of oral antihyperglycemic agents, pentoxifylline and/or theophylline;
  9. Use of any drug therapy that directly affects gastrointestinal motility;
  10. History of any significant drug allergy;
  11. History of difficulty with phlebotomy;
  12. Use of any recreational drugs within the past year or a previous history of drug or alcohol abuse;
  13. Positive results from a urine screen for alcohol or substances of abuse at screening or upon admission to the Clinic;
  14. Current smoker or user of any tobacco products;
  15. Use of any prescription drug therapy within 14 days prior to receiving study drug, with the exception of therapy to treat DM;
  16. Use of any over-the-counter (OTC) drugs or herbal preparations within 72 hours prior to receiving study drug;
  17. Consumption of any caffeine-containing foods or beverages within 24 hours prior to receiving study drug;
  18. Consumption of alcohol within 24 hours prior to admission to the Clinic;
  19. Consumption of any grapefruit or grapefruit-containing juices within 72 hours prior to receiving study drug;
  20. Use of an investigational drug or product, or participation in a drug research study within 30 days prior to receiving drug;
  21. Prior exposure to lisofylline;
  22. The donation of blood (1 pint or more) within 30 days or plasma within 7 days of receiving study drug;
  23. Any condition which in the opinion of Investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he or she took part in the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety (based on AEs, vital signs assessments, resting 12-lead ECG evaluations, physical examination findings and clinical laboratory test results) | LSF Plasma levels: D1-2, 7-8; T 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24 h; D2, 8; T 5, 10, 15, 30 min and 1, 2, 3, 4, 6, 8, 10, 12, 16 h post inf. Cytokine, chemokine, insulin, free fatty acid STAT4 phosphorylation in monocytes: D1-2, 7-8

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters will include AUC0-t, AUC0-inf, Cmax, Tmax, t1/2, kel, CL, Vdss and F | LSF Plasma levels: D1-2, 7-8; T 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24 h; D2, 8; T 5, 10, 15, 30 min and 1, 2, 3, 4, 6, 8, 10, 12, 16 h post inf. Cytokine, chemokine, insulin, free fatty acid STAT4 phosphorylation in monocytes: D1-2, 7-8
Pharmacodynamic (PD) assessments (blood will be collected for determination of serum cytokine, chemokine, insulin and FFA levels at time points noted previously) | LSF Plasma levels: D1-2, 7-8; T 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24 h; D2, 8; T 5, 10, 15, 30 min and 1, 2, 3, 4, 6, 8, 10, 12, 16 h post inf. Cytokine, chemokine, insulin, free fatty acid STAT4 phosphorylation in monocytes: D1-2, 7-8

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Biomedical Research, Inc. (ABR), Hackensack, New Jersey, United States